CLINICAL TRIAL: NCT05042271
Title: Pharmacokinetics of Meropenem in Patients on Plasma Exchange
Brief Title: PK of Meropenem in Patients on Plasma Exchange
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Sutep Jaruratanasirikul, Department of Internal Medicine, Faculty of Medicine, Prince of Songkla University, Prince of Songkla University
Other Study IDs: meropenem-plasma exchange
Record Dates: First submitted 2021-07-13; First posted 2021-09-13 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Autoimmune Diseases
Keywords: therapeutic plasma exchange; meropenem; pharmacokinetic
MeSH Terms: conditions — Autoimmune Diseases | interventions — Meropenem

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Meropenem: Patients who underwent TPE (Phase 1): In phase 1, each patient received a 1 hour infusion of a single dose of 1 g of meropenem diluted in 100 ml of normal saline solution, at the same time as the start of the first therapeutic plasma exchange (TPE) and meropenem PK studies were carried out after the administration of meropenem. Blood samples (3 ml) were obtained by direct venipuncture at the following times: shortly before (time zero) and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6 and 8 hours after the start of the meropenem administration.
  Interventions: Drug: meropenem
- Meropenem: after TPE (Phase 2): was similar to phase 1 except that the meropenem administration and PK studies were conducted >6 hours apart from the next TPE
  Interventions: Drug: meropenem

INTERVENTIONS:
Drug: meropenem — each patient received a 1 hour infusion of a single dose of 1 g of meropenem diluted in 100 ml of normal saline solution, at the same time as the start of the first TPE and meropenem PK studies were carried out after the administration of meropenem. Blood samples (3 ml) were obtained by direct venipuncture at the following times: shortly before (time zero) and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6 and 8 hours after the start of the meropenem administration.

SUMMARY:
Therapeutic plasma exchange (TPE) has been shown to be an important procedure for treatment of a variety of refractory immune complex disorders, such as Guillain-Barré syndrome and neuromyelitis optica. The intervention removes plasma, albumin, or some other substance. Meropenem is a broad-spectrum beta-lactam antimicrobial agent that is used for the treatment of serious nosocomial infections. Pathophysiological changes in patients on TPE can alter the pharmacokinetic (PK) patterns of coadministered antibiotics. This effect has an impact on the antimicrobial agents when paticipants are administered during the intervention. The aim of this study was to investigate the impact of TPE on meropenem PK.

ELIGIBILITY:
Inclusion Criteria:

* age≥ 18 years
* no shock
* hemoglobin ≥ 7 g/dl

Exclusion Criteria:

* pregnancy or breast-feeding female
* history of hypersensitivity to carbapenems
* renal replacement therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: autoimmune diseases
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-10-18 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The plasma concentrations were measured at the following times: 0, 0.25, 0.5, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6 and 8 hour after the start of drug administration | 0-8 hours after the drug administration

SECONDARY OUTCOMES:
Maximum plasma concentration [Cmax] | 0-8 hours after the drug administration
Minimum plasma concentration [Cmin] | 0-8 hours after the drug administration
Area under the plasma concentration versus time curve [AUC] | 0-8 hours after the drug administration
half-life [t1/2] | 0-8 hours after the drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Sutep Jaruratanasirikul, M.D., Principal Investigator — Faculty of Medicine, Prince of Songkla University, Thailand
Locations (1):
- Faculty of Medicine, Prince of Songkla University, Thailand, Hat Yai, Changwat Songkhla, Thailand